CLINICAL TRIAL: NCT01319305
Title: BREATHE Long-Term Follow-Up Study
Status: Completed | Type: Observational
Sponsor: Entellus Medical, Inc. (Industry)
Responsible Party: Robyn Schacherer, Principal CRA, Entellus Medical
Other Study IDs: 1743-001
Record Dates: First submitted 2011-03-14; First posted 2011-03-21 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Sinus Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BREATHE I participatants
  Interventions: Device: FinESS Sinus Treatment

INTERVENTIONS:
Device: FinESS Sinus Treatment — balloon sinuplasty

SUMMARY:
This is a long-term follow-up of patients that participated in the BREATHE I study.

ELIGIBILITY:
Inclusion Criteria:

* Participated in BREATHE I study
* Willing to sign consent and participate in long-term follow-up study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who were treated with FinESS Sinus Treatment in the BREATHE I Study
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
SNOT-20 scores | approximately 24 months
  Assess post-procedure outcomes defined as SNOT-20 scores and work productivity assessment questionnaires aproximately 24 months post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- St. Cloud ENT, Saint Cloud, Minnesota, United States